CLINICAL TRIAL: NCT00625989
Title: The Effect of Allergen Inhalation on Sputum Myeloid and Plasmacytoid Dendritic Cells in Mild Atopic Asthmatics
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: sputdend08; BDUA2008
Record Dates: First submitted 2008-01-23; First posted 2008-02-29 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2015-04

CONDITIONS: Asthma
Keywords: asthma; atopy; allergen challenge; sputum myeloid and plasmacytoid dendritic cells
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diluent (Placebo Comparator): Inhalation challenge preformed with diluent.
  Interventions: Drug: Aeroallergen
- Allergen (Active Comparator): Inhalation challenge preformed with allergen.
  Interventions: Drug: Aeroallergen

INTERVENTIONS:
Drug: Aeroallergen

SUMMARY:
Summary:

A picture is emerging of dendritic cells migrating through the blood to the airways following allergen inhalation in atopic asthmatics. Although the Koh and McCarthy articles present novel findings, both do not provide a comprehensive view of sputum DCs following allergen challenge. Therefore, the proposed study will examine the kinetics of mDCs and pDCs in the induced sputum of atopic asthmatics following inhalation of allergen.

Hypothesis:

Following allergen challenge, sputum myeloid and plasmacytoid DCs will migrate into the airway lumen in atopic asthmatics during the timeframe of the late asthmatic response.

Objective:

The objective of this study is to examine the kinetics of dendritic cells in induced sputum following allergen challenge in atopic asthmatic subjects.

DETAILED DESCRIPTION:
Subjects will be put through two study periods. Each study period will consist of four visits and will be separated by 2-4 weeks. On the first visit, subjects will undergo screening procedures, including complete history and physical examination. In addition, methacholine inhalation challenge and skin-prick testing will be preformed to assess airway hyper-responsiveness and determine atopic status respectively. Lastly, sputum will be induced before challenge (0 hrs) and peripheral blood will be collected. On the second visit, subjects will inhale diluent or allergen and sputum will be collected 7 hours following inhalation challenge. Next, on the third visit, subjects will return 24 hours following inhalation challenge and sputum will be induced. On the final visit, subjects will return 72 hours following inhalation challenge and sputum will be collected, along with peripheral blood.

Before the next study period begins, there will be a washout period of 2-4 weeks. On the first visit of the second study period, a methacholine challenge will be performed to ensure the return of PC20 to within one doubling dose of baseline values. Also, sputum will be induced before challenge (0hrs) and peripheral blood will be collected. On the second visit, subjects will inhale diluent or allergen and sputum will be collected 7hrs following inhalation challenge. Next, on the third visit, subjects will return 24 hours following inhalation challenge and sputum will be induced. On the final visit, subjects will return 72 hours following inhalation challenge and sputum will be collected, along with peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Mild atopic asthmatics, presently well controlled on ß2-agonists.
* Non-smokers.
* Baseline FEV1 more than 70% of predicted normal.

Exclusion Criteria:

* Airway infection during the last 4 weeks.
* Exacerbation during the last 4 weeks.
* Inhaled or oral steroids during the last 4 weeks.
* Antihistamines during the last 48 hours.
* Asthma medication other than inhaled and/or oral ß2-agonists during the last 4 weeks.
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Principal Investigator — McMaster University; Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Diluent Then Allergen Challenge: Subjects were screened, then given a 2 week washout period.
  Samples collected on day 1 according to protocol. Day 2 diluent challenge was preformed and samples collected according to the protocol. Subjects returned on day 3 for 24 hour follow up and samples collected according to the protocol.
  Two week wash out period.
  Samples collected on day 1, after washout, according to protocol. Day 2, after washout, allergen challenge was preformed and samples collected according to the protocol. Subjects returned on day 3, after wash out, for 24 hour follow up and samples collected according to the protocol.
- Allergen Then Diluent Challenge: Subjects were screened, then given a 2 week washout period.
  Samples collected on day 1 according to protocol. Day 2 allergen challenge was preformed and samples collected according to the protocol. Subjects returned on day 3 for 24 hour follow up and samples collected according to the protocol.
  Two week wash out period.
  Samples collected on day 1, after washout, according to protocol. Day 2, after washout, dilluent challenge was preformed and samples collected according to the protocol. Subjects returned on day 3, after wash out, for 24 hour follow up and samples collected according to the protocol.
Period: Overall Study
Arm/Group | Diluent Then Allergen Challenge | Allergen Then Diluent Challenge
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mild Asthmatics: Mild asthmatics who require only short-acting beta agonist bronchodilator treatment as required.
Arm/Group | Mild Asthmatics
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure for This Study is the Number of Sputum Myeloid Dendritic Cells
Description: Flow-cytometric acquisitions were used to determine the percentage of each type of mononuclear cell. These percentages were multiplied by the number of sputum mononuclear cells calculated by using total and differential cell counts of the sputum sample.
Time Frame: 24 hrs
Measure: Mean (Standard Deviation); unit: number of cells/g of sputum
Groups:
- Diluent; Allergen: Mild asthmatics who require only short-acting beta agonist bronchodilator treatment as required.
Arm/Group | Diluent | Allergen
Number analyzed (Participants) | 12 | 12
number of cells/g of sputum | 32800 (13100) | 89100 (27000)

2. Primary Outcome: The Primary Outcome Measure for This Study is the Number of Sputum Plasmacytoid Dendritic Cells
Description: as for outcome 1
Time Frame: 24 hrs
Measure: Mean (Standard Deviation); unit: number of cells/g of sputum
Arm/Group | Diluent | Allergen
Number analyzed (Participants) | 12 | 12
number of cells/g of sputum | 16000 (8700) | 39900 (12200)

3. Secondary Outcome: The Secondary Outcome Measure is the Level of Specific Chemokines Released in the Sputum Supernatant.
Time Frame: Before inhalation (0hrs)
Reporting Status: Not Posted

4. Secondary Outcome: The Secondary Outcome Measure is the Level of Specific Chemokines Released in the Sputum Supernatant
Time Frame: 7 hrs
Reporting Status: Not Posted

5. Secondary Outcome: The Secondary Outcome Measure is the Level of Specific Chemokines Released in the Sputum Supernatant
Time Frame: 24 hrs
Reporting Status: Not Posted

6. Secondary Outcome: The Secondary Outcome Measure is the Level of Specific Chemokines Released in the Sputum Supernatant
Time Frame: 72 hrs
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Mild Asthmatics
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes